CLINICAL TRIAL: NCT02947451
Title: Immediate Effects of Manual Therapy Versus TENS in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriel Peixoto Leão Almeida (Other)
Responsible Party: Sponsor-Investigator, Gabriel Peixoto Leão Almeida, Master, Universidade Federal do Ceara
Organization: Universidade Federal do Ceara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TCC_Isabel
Record Dates: First submitted 2016-09-06; First posted 2016-10-27 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Musculoskeletal Manipulations; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual therapy (Experimental): In manual therapy group will be assigned a protocol with manual passive stretching for the quadriceps muscles, hamstrings, triceps surae, adductors and abductors of the hip; myofascial release peripatellar; joint mobilization grades 1 and 2 for tibiofemoral joint and femoro - patellar in the affected knee, in a single application.
  Interventions: Other: Manual Therapy
- TENS (Experimental): In TENS group will be applied to continuous current mode, frequency 100Hz and pulse width of 50μs for 40 minutes in a single application.
  Interventions: Other: TENS

INTERVENTIONS:
Other: Manual Therapy — In manual therapy group will be assigned a protocol with manual passive stretching for the quadriceps muscles, hamstrings, triceps surae, adductors and abductors of the hip; myofascial release peripatellar; joint mobilization grades 1 and 2 for tibiofemoral joint and femoro - patellar in the affected knee.
  Stretching, myofascial release and mobilizations will be held for 30 seconds, with three repetitions of each. The intervention will be applied only once.
  Arms: Manual therapy
Other: TENS — In TENS group will be applied to continuous current mode, frequency 100Hz and pulse width of 50μs for 40 minutes in a single application. The intensity will be defined by the patient, should the stimulus be considered intense, but pleasant to it.
  Other Names: Transcutaneous electrical nerve stimulation
  Arms: TENS

SUMMARY:
Patients with knee Osteoarthritis have high prevalence of pain , requiring ever more precise interventions in their management. This study aims to investigate the immediate effects of manual therapy and TENS on pain in patients with knee Osteoarthritis. Knowledge of best interventions favors reducing spending on health and safety for the patient.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of manual therapy and TENS for immediate control of pain in patients with knee osteoarthritis. They will be included 62 patients with clinical and radiological diagnosis of knee osteoarthritis, presenting pain of at least 3 in VAS, which are recruited from rheumatology and geriatrics clinics in Fortaleza / CE through a prior screening.

Will be three assessments, prior to the intervention, immediately after it and after 72 hours. The data collected shall appear in individual printed records. Participants will be divided into two therapy groups, of which one will be applied manual therapy and other TENS. There will be randomisation allocation of individuals in the groups and because of the nature of the interventions only the evaluator may be blind.

In manual therapy group will be assigned a protocol with manual passive stretching for the quadriceps muscles, hamstrings, triceps surae, adductors and abductors of the hip; myofascial release peripatellar; joint mobilization grades 1 and 2 for tibiofemoral joint and femoro - patellar in the affected knee.

In TENS group will be applied to continuous current mode, frequency 100Hz and pulse width of 50μs for 40 minutes in a single application. The intensity will be defined by the patient, should the stimulus be considered intense, but pleasant to it.

The Kolmogorov - Smirnov test is used to verify the data distribution normality. The characterization of the participants is performed by means of descriptive statistical analysis. Parametric or non-parametric tests will be used according to the data distribution normality for comparison between groups at baseline. The evaluator blinding will be tested using the chi -square test by comparing the randomization code with the evaluator opinion. The difference between the groups and their respective confidence intervals will be calculated by linear mixed models using interaction term of "time versus group."

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis diagnosed by clinical criteria established by the American College of Rheumatology and radiological criteria of Kelgren-Lawrence
* Age over 50 years
* Pain intensity above 2 on the VAS

Exclusion Criteria:

* Other systemic inflammatory disease
* Changes in sensitivity
* Use of anti-inflammatory steroids, tranquillizers and/or antidepressants in the last month
* Analgesic in last 24 hours
* Use of cardiac pacemaker

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity in Visual Analogic Scale | Immediately
  It consists of 11 points, ranging from 0 ( no pain) to 10 ( maximum possible pain ), the volunteer instructed to quantify their knee pain present at the time of evaluation.
Pressure Pain Threshold in Algometer | Immediately
  They will be scored 7 points, the first being located at the apex of the patella, the second three cm medial to the apex of the patella, the third two centimeters higher than the second, the fourth two centimeters lower than the second, the fifth three centimeters lateral to the apex of the patella, the sixth two centimeters above the fifth and seventh two centimeters below the fifth.
  Participants will be instructed to report to the appraiser whenever the feeling in the stimulus site becomes clearly painful. There will be two measurements at each point, each starting from point 1 to 7. It shall be considered the average of each isolated point and the average of the averages of the points how test result.

SECONDARY OUTCOMES:
Global Rating of Change Scale | Immediately and 72 hours after intervention
  Used to evaluate the self- perception of the volunteer about the overall state of the affected knee. It is formed by 11 points, ranging from -5 (much worse), 0 (unchanged) to +5 (completely better), the participant instructed to quantify their perception with the question: "Compared to their condition before the treatment, how would you describe your knee right now?"
Pain intensity in Visual Analogic Scale 72 hours after intervention | 72 hours after intervention
  It consists of 11 points, ranging from 0 ( no pain) to 10 ( maximum possible pain ), the volunteer instructed to quantify their knee pain present at the time of evaluation.
Pressure Pain Threshold in Algometer 72 hours after intervention | 72 hours after intervention
  They will be scored 7 points, the first being located at the apex of the patella, the second three cm medial to the apex of the patella, the third two centimeters higher than the second, the fourth two centimeters lower than the second, the fifth three centimeters lateral to the apex of the patella, the sixth two centimeters above the fifth and seventh two centimeters below the fifth.
  Participants will be instructed to report to the appraiser whenever the feeling in the stimulus site becomes clearly painful. There will be two measurements at each point, each starting from point 1 to 7. It shall be considered the average of each isolated point and the average of the averages of the points how test result.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedson J, Jordan K, Croft P. The prevalence and history of knee osteoarthritis in general practice: a case-control study. Fam Pract. 2005 Feb;22(1):103-8. doi: 10.1093/fampra/cmh700. Epub 2005 Jan 7. PMID 15640302
- [Background] Deyle GD, Gill NW, Allison SC, Hando BR, Rochino DA. Knee OA: which patients are unlikely to benefit from manual PT and exercise? J Fam Pract. 2012 Jan;61(1):E1-8. PMID 22220299
- [Background] Alshami AM. Knee osteoarthritis related pain: a narrative review of diagnosis and treatment. Int J Health Sci (Qassim). 2014 Jan;8(1):85-104. doi: 10.12816/0006075. PMID 24899883
- [Background] French HP, Brennan A, White B, Cusack T. Manual therapy for osteoarthritis of the hip or knee - a systematic review. Man Ther. 2011 Apr;16(2):109-17. doi: 10.1016/j.math.2010.10.011. Epub 2010 Dec 13. PMID 21146444
- [Background] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Abbott JH, Robertson MC, Chapple C, Pinto D, Wright AA, Leon de la Barra S, Baxter GD, Theis JC, Campbell AJ; MOA Trial team. Manual therapy, exercise therapy, or both, in addition to usual care, for osteoarthritis of the hip or knee: a randomized controlled trial. 1: clinical effectiveness. Osteoarthritis Cartilage. 2013 Apr;21(4):525-34. doi: 10.1016/j.joca.2012.12.014. Epub 2013 Jan 8. PMID 23313532
- [Background] Brantingham JW, Bonnefin D, Perle SM, Cassa TK, Globe G, Pribicevic M, Hicks M, Korporaal C. Manipulative therapy for lower extremity conditions: update of a literature review. J Manipulative Physiol Ther. 2012 Feb;35(2):127-66. doi: 10.1016/j.jmpt.2012.01.001. PMID 22325966
- [Background] Jansen MJ, Viechtbauer W, Lenssen AF, Hendriks EJ, de Bie RA. Strength training alone, exercise therapy alone, and exercise therapy with passive manual mobilisation each reduce pain and disability in people with knee osteoarthritis: a systematic review. J Physiother. 2011;57(1):11-20. doi: 10.1016/S1836-9553(11)70002-9. PMID 21402325
- [Background] Moss P, Sluka K, Wright A. The initial effects of knee joint mobilization on osteoarthritic hyperalgesia. Man Ther. 2007 May;12(2):109-18. doi: 10.1016/j.math.2006.02.009. Epub 2006 Jun 13. PMID 16777467
- [Background] Pollard H, Ward G, Hoskins W, Hardy K. The effect of a manual therapy knee protocol on osteoarthritic knee pain: a randomised controlled trial. J Can Chiropr Assoc. 2008 Dec;52(4):229-42. PMID 19066697
- [Background] Basedow M, Williams H, Shanahan EM, Runciman WB, Esterman A. Australian GP management of osteoarthritis following the release of the RACGP guideline for the non-surgical management of hip and knee osteoarthritis. BMC Res Notes. 2015 Oct 5;8:536. doi: 10.1186/s13104-015-1531-z. PMID 26438323
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Bjordal JM, Johnson MI, Lopes-Martins RA, Bogen B, Chow R, Ljunggren AE. Short-term efficacy of physical interventions in osteoarthritic knee pain. A systematic review and meta-analysis of randomised placebo-controlled trials. BMC Musculoskelet Disord. 2007 Jun 22;8:51. doi: 10.1186/1471-2474-8-51. PMID 17587446
- [Background] Nnoaham KE, Kumbang J. WITHDRAWN: Transcutaneous electrical nerve stimulation (TENS) for chronic pain. Cochrane Database Syst Rev. 2014 Jul 10;(7):CD003222. doi: 10.1002/14651858.CD003222.pub3. No abstract available. PMID 25010718
- [Background] Vance CG, Rakel BA, Blodgett NP, DeSantana JM, Amendola A, Zimmerman MB, Walsh DM, Sluka KA. Effects of transcutaneous electrical nerve stimulation on pain, pain sensitivity, and function in people with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2012 Jul;92(7):898-910. doi: 10.2522/ptj.20110183. Epub 2012 Mar 30. PMID 22466027
- [Background] Mascarin NC, Vancini RL, Andrade ML, Magalhaes Ede P, de Lira CA, Coimbra IB. Effects of kinesiotherapy, ultrasound and electrotherapy in management of bilateral knee osteoarthritis: prospective clinical trial. BMC Musculoskelet Disord. 2012 Sep 22;13:182. doi: 10.1186/1471-2474-13-182. PMID 22999098
- [Background] Bellamy N. Osteoarthritis clinical trials: candidate variables and clinimetric properties. J Rheumatol. 1997 Apr;24(4):768-78. PMID 9101516
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Roos EM, Roos HP, Ekdahl C, Lohmander LS. Knee injury and Osteoarthritis Outcome Score (KOOS)--validation of a Swedish version. Scand J Med Sci Sports. 1998 Dec;8(6):439-48. doi: 10.1111/j.1600-0838.1998.tb00465.x. PMID 9863983
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Cheing GL, Tsui AY, Lo SK, Hui-Chan CW. Optimal stimulation duration of tens in the management of osteoarthritic knee pain. J Rehabil Med. 2003 Mar;35(2):62-8. doi: 10.1080/16501970306116. PMID 12691335
- [Background] Law PP, Cheing GL. Optimal stimulation frequency of transcutaneous electrical nerve stimulation on people with knee osteoarthritis. J Rehabil Med. 2004 Sep;36(5):220-5. doi: 10.1080/16501970410029834. PMID 15626162